CLINICAL TRIAL: NCT03031288
Title: Vented Base Feeding Bottle in Preterm Infants With GERD Symptoms: Effects on Respiration-swallow Patterns and Reflux.
Brief Title: Effects of Vented Base Feeding Bottle in Preterm Infants With GERD Symptoms.
Acronym: FeedGERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Cresi, MD, PhD, MD PhD, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: feeding-01
Record Dates: First submitted 2017-01-12; First posted 2017-01-25 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: GERD; Apnea Neonatal
Keywords: gastroesophageal reflux; swallow; feeding bottle; cardiorespiratory; apnoea; preterm; impedance-pH-metry
MeSH Terms: conditions — Gastroesophageal Reflux; Bottle Feeding; Apnea; Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Start feeding with Device A, "standard" (Experimental): Alternatively feeding with standard feeding bottle (Device A) and vented base feeding bottle (Device B)
  Interventions: Device: A; Device: B
- Start feeding with Device B, "vented" (Experimental): Alternatively feeding with vented base feeding bottle (Device B) and standard feeding bottle (Device A)
  Interventions: Device: A; Device: B

INTERVENTIONS:
Device: A — standard bottle
Device: B — vented base bottle

SUMMARY:
Aim of the study is to evaluate the effects of vented base bottles on respiration-swallow patterns and on gastroesophageal refluxes in preterm infants with clinical suspect of gastroesophageal reflux disease (GERD).

In this crossover-randomized study, we compared the effects of standard feeding bottles (A) versus vented base feeding bottles (B) on a group of patients with at least 2 clinical GERD symptoms. 24 hours of synchronized cardiorespiratory (CR) and Esophageal Multichannel intraluminal impedance (MII/pH) monitoring were evaluated for each patient. During this period, patients were fed alternatively with feeding bottle A and B.

DETAILED DESCRIPTION:
In preterm infants a deficit of both coordination and gastro-intestinal motility is often the underpinning cause of oxygen desaturations and gastro-esophageal reflux. Breastfeeding enhances the maturation of the respiration-swallow mechanism. For this reason, a feeding bottle that best recreates the physiological sucking from the maternal breast is highly desirable in non-breastfed newborns.

Population: newborns referred to esophageal Multichannel Intraluminal Impedance and pH-metry (MII/pH) combined with cardiorespiratory (CR) monitoring for GERD or cardio-respiratory symptoms

Materials and methods: we compare the effects of traditional feeding bottles (A) versus vented base feeding bottles (B) on cardiorespiratory and reflux events in newborns undergoing 24 hours synchronized CR and MII/pH monitoring. During the exam, newborns are fed, alternatively, by feeding bottle A and B with human milk or formula. Some training meals are offered the day before monitoring to get newborns enrolled into the study used to vented base feeding bottles.

Cardiorespiratory monitoring is performed through VitaGuard VG3100® (Getemed Medizin- und Informationstechnik AG, Teltow, Germany) based on Masimo Signal Extraction Technology (SET)® (Masimo Corp., Irvine, CA, USA). It operates with a blood oxygen saturation (SpO2) detector, placed on the right wrist, and 3 thoracic electrodes. This instrument is able to record ECG, heart rate, SpO2 and thoracic plethysmographic curve. The signals are analyzed with VitaWin 3® software (Getemed Medizin - und Informationstechnik AG, Teltow, Germany), by filtering artifacts.

The MII/pH monitoring is performed through a neonatal catheter (Infant Comfort TEC®) with 7 impedence electrodes (creating 6 impedance channels) and one pH detector able to cover the whole distance from the pharynx to the lower esophageal sphincter (LES) (channel 1). The pH detector is placed within channel 1, 1.5 cm above the LES. The correct positioning of the catheter is measured through fluoroscopy and eventually corrected. Data obtained from impedance channels that result proximal to the superior esophageal sphincter are excluded from the analysis. The acquisition and recording of MII/pH data are performed through Sleuth System, Sandhill Scientific Inc., Highlands Ranch, Colorado, USA. The analysis of MII/pH tracings is made visually by a single operator using BioView 5.3.4 software (Sleuth System, Sandhill Scientific Inc., Highlands Ranch, Colorado, USA).

The variables analyzed are listed as follows:

Clinical variables:

* feeding time (min)
* feeding total volume (mL)
* n. GER during feeding
* n. GER in the post-prandial period (150 min after feeding)

Cardiorespiratory variables:

* frequency of apnea, desaturation and bradycardia during feeding
* frequency of apnea, desaturation and bradycardia during post-prandial period
* mean duration of apnea during feeding and post-prandial period
* mean and minimum desaturation level during feeding and post-prandial period
* mean and minimum heart rate during feeding and post-prandial period

MII/pH variables:

* Swallow frequency during feeding and post-prandial period (events/h)
* Bolus Presence Time (BPT): seconds between bolus entry and bolus exit in the distal channel
* Bolus Head Advancing Time (BHAT): seconds between bolus entry in proximal channel and entry in distal channel
* Bolus Head Advancing Time Corrected for Esophageal Length (BHATc): BHAT corrected for esophageal length (BHATc = BHAT / esophageal length)
* Reflux pH: minimum pH value registered during each GER event. It classifies refluxes into 3 different types: acid (pH < 4), weakly acid (pH 4-7) and weakly alkaline (pH > 7)
* GER frequency, (events/h)
* Bolus Clearance Time (BCT): reflux duration, recorded at distal channel (s)
* Bolus Reflux Extent (BRE), (n. channels)
* Proximal GER frequency (events/h)
* Bolus Exposure Index (BEI): percentage of time in which GER involves esophagus during MII/pH monitoring
* Reflux Index (RI): percentage of time during which pH falls below 4 during MII/pH monitoring

Randomization: the alternate use of feeding bottles A and B is set by a binary random sequencing generated by Microsoft Office Excel software that indicates the first feeding bottle to be used. This is a single-blind study since the sequence is unknown to the specialist in charge of reporting MII/pH and CR monitoring.

Statistical analysis:

The analysis is made with Statistical Software Package For Windows® (StatSoft, Inc., Tulsa, Oklahoma, USA). Kolmogorov-Smirnov test and exploratory data analysis are used to define normality range. Data will be expressed as mean and standard deviation (SD), or as median and interquartile range if more appropriate. Differences among cardiorespiratory and MII/pH variables will be evaluated with Student paired T test or Wilcoxon test if more appropriate. Significance will be considered as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* weight ≥ 1500 g at the time of examination
* at least 2 GERD symptoms
* exclusive enteral feeding
* parents' informed consent

Exclusion Criteria:

* congenital abnormalities
* perinatal asphyxia
* respiratory, genetic, metabolic, infectious and/or neurologic disease
* pharmacological therapies, in the last 7 days, able to affect esophageal motility

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Frequency of cardiorespiratory events (feeding+postprandial time) | calculated throughout 24 hour
  Cardiorespiratory events / hour
  * apnea (no breathing movement for at least 20 s, or less if associated with desaturation/bradycardia)
  * desaturation (SpO2 <80%)
  * bradycardia (heart rate < 80 bpm for at least 1 s)

SECONDARY OUTCOMES:
Swallow event characteristics (feeding time) | calculated throughout 30 minute interval after the beginning of the milk meal
  Swallow event is identified as a rapid increase in impedance preceded by a drop in impedance to 50% of baseline beginning in the proximal channel and proceeding in an anterograde direction to the most distal channel, followed by the recovery of baseline values at each channel
Frequency of reflux events (postprandial time) | calculated throughout 150 minute interval after the end of the milk meal
  Reflux event is defined as: a drop of impedance to 50% of the basal value for at least 5 s, starting in the most distal channel and proceeding to one or more proximal channels and followed by a recovery of the impedance baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, MD PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- Ospedale S.Anna di Torino, Torino, (TO), Italy

IPD SHARING:
Plan to Share IPD: No